CLINICAL TRIAL: NCT04961333
Title: Internet-based Multidisciplinary Rehabilitation for Longterm COVID-19 Syndrome
Acronym: COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danderyd Hospital (Other)
Collaborators: St Göran Hospital, Stockholm (Unknown)
Responsible Party: Principal Investigator, Indre Ljungar, associated professor in rehabilitation medicine, Danderyd Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Danderyd University Hospital
Record Dates: First submitted 2021-05-07; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Long COVID-19
Keywords: COVID-19; rehabilitation; telemedicine; multidisciplinary
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: Intervention group and waiting list control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation group (Experimental): Rehabilitation group will be provided multidisciplinary interventions online and individually by ExorLive app. The screening with self-scored questionnaires and physical tests will be performed before and after 8 weeks rehabilitation.
  Interventions: Behavioral: Multidisciplinary Rehabilitation
- Waiting list controls (No Intervention): Passive waiting list or control group, which will be offered to participate in rehabilitation after at least 8 weeks of waiting time. The group will fulfil screening twice, following the time schedule of intervention group. When invited to rehabilitation a new screening will be asked to be completed if the waiting time after the last screening will be longer than 2 weeks.

INTERVENTIONS:
Behavioral: Multidisciplinary Rehabilitation — Body therapies to improve breathing, normalise dysfunction in the autonomic nervous system, relaxation, mindfulness, in some part Acceptance and Commitment Therapy given preferably through body therapies.
  Other Names: Individually performed physical activity recorded into ExorLie app.
  Arms: Rehabilitation group

SUMMARY:
Internet-based multidisciplinary interventions will be offered to participants suffering from longterm COVID-19 syndrome. Data will be collected by internet platform at Karolinska Institutet (BASS) before, after rehabilitation and at follow-up after 6 months. Both self-scored questionnaires and physical tests performed at home will be collected to understand the symptomatology, functioning and activity level. Rehabilitation during 8 weeks period will be given in groups as face-to-group, pre-recorded film sessions and by individual approach, the participants will use ExorLive app for physical activity.

DETAILED DESCRIPTION:
This randomised study aimed to understand if multidisciplinary internet-based interventions performed in group and individually are applicable for participants suffering from longterm COVID-19 syndrome. Data will be collected by internet platform at Karolinska Institutet (BASS) before, after rehabilitation and at follow-up after 6 months. Both self-scored questionnaires and physical tests performed at home will be collected to understand the symptomatology, functioning and activity level. Rehabilitation during 8 weeks period will be given in groups as face-to-group, pre-recorded film sessions and by individual approach, the participants will use ExorLive app for physical activity.

The participants will be randomised for treatment and waiting lists using a website random.org. Waiting list will be offered rehabilitation interventions after at least 8 weeks period of waiting to exclude a spontaneous improvement or worsening of symptoms. To understand the impact of rehabilitation on work capacity and employment/economic supply, the data from Social Insurance databas will be obtained 2021 year before and upp to 2 years after the intervention. To understand the impact of rehabilitation on sickness-leave, the data from National Insurance Agency will be obtained for 2021 and 2022.

ELIGIBILITY:
Inclusion Criteria:

* confirmed COVID-19 infection
* post-infection symptoms lasting longer than 3-6 months
* clinically stable persons regarding symtoms or other co-morbidities
* ability to participate in internet-based rehabilitation in group in Swedish.

Exclusion Criteria:

* uncertainty regarding covid-19 infection or co-morbidities started or exacerbated during the same time
* alcohol and drug abuse
* untreated psychiatric and somatic co-morbidities
* undergoing medical or psychotherapeutic treatment or rehabilitation which can interact with rehabilitation outcomes.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in health-related quality of life measured by Short Form-36 | Investigators expect changes at 6 months follow-up after rehabilitation
  Important sub scales: vitality, general health, physical functioning, pain. Scale varies between 0 and 100 (highest)
Changes in heart rate variability during physical tests | Investigators expect normalisation at 6 months follow-up
  Heart rate variability measured by puls oximeter during 2 physical tests

SECONDARY OUTCOMES:
Overall changed scores in validated questionnaires for fatigue, breathing, pain and sleep disorders | Investigators expect changes already at 6 months follow-up
  Validated self-scored questionnaires such as Multidimentional Fatigue Inventory - for fatigue (values 0-20), Clinical COPD Questionnaire - for breathing (0-50), Chronic Visual Analogue Scale - for pain (0-100), Insomnia Severity Scale - for sleep (0-21) and other questionnaires.
Changed functioning and activity | Investigators expect normalisation at 6 months follow-up
  Functioning and activity will be evaluated by self-scored questionnaires and a new questionnaire Functional compass for COVID-19 based on ICF (International Classification of Functioning and Disability)

CONTACTS AND LOCATIONS:
Locations (1):
- St Göran Hospital, Stockholm, Sweden